CLINICAL TRIAL: NCT00028717
Title: A Randomized Phase III Study Of Chimeric Anti-CD20 Monoclonal Antibody (Rituximab) With 2-Weekly CHOP Chemotherapy In Elderly Patients With Intermediate Or High-Risk Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy Plus Filgrastim With or Without Rituximab in Treating Older Patients With Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Commissie Voor Klinisch Toegepast Onderzoek (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000069122; CKTO-2000-10; HOVON-46NHL; EU-20130; HOVON-CKVO-2000-10
Record Dates: First submitted 2002-01-04; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-11

CONDITIONS: Lymphoma
Keywords: stage I grade 3 follicular lymphoma; stage I adult diffuse large cell lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse large cell lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — Filgrastim; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells. It is not yet known if combination chemotherapy plus filgrastim is more effective with or without rituximab in treating non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to determine the effectiveness of combination chemotherapy plus filgrastim with or without rituximab in treating older patients who have non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of cyclophosphamide, doxorubicin, vincristine, prednisone (CHOP), and filgrastim (G-CSF) with or without rituximab on event-free survival of elderly patients with intermediate or high-risk non-Hodgkin's lymphoma.
* Compare the complete remission rate, overall survival, and disease-free survival of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, WHO classification, and International Prognostic Index score. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1; oral prednisone on days 1-5; and filgrastim (G-CSF) subcutaneously on days 1-14. Treatment repeats every 2 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive cyclophosphamide, doxorubicin, vincristine, prednisone, and G-CSF as in arm I. Patients also receive rituximab IV on day 3 of courses 1-2 and on day 1 of courses 3-6 for a total of 6 doses.

Patients are followed every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 400 patients (200 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-Hodgkin's lymphoma (NHL)

  * Low- or high-intermediate or high-risk lymphoma of any of the following subtypes:

    * Mantle cell lymphoma
    * Follicular lymphoma (grade III)
    * Diffuse large B-cell lymphoma
* CD20-positive
* No suspected or documented CNS involvement by NHL NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 65 and over

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 1.75 mg/dL*
* Transaminases less than 2.5 times normal* NOTE: * Unless due to NHL

Renal:

* Creatinine less than 1.7 mg/dL (unless due to NHL)

Cardiovascular:

* No severe cardiac dysfunction
* No New York Heart Association class II-IV heart disease
* LVEF at least 45%

Pulmonary:

* No uncontrolled asthma requiring steroid treatment

Other:

* HIV negative
* No intolerance to exogenous protein administration
* No active, uncontrolled infection
* No uncontrolled allergy requiring steroid treatment
* No other malignancy within the past 5 years except basal cell skin cancer or stage 0 cervical cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy for NHL

Chemotherapy:

* No prior chemotherapy for NHL

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy for NHL except local radiotherapy for potential organ dysfunction by localized lymphoma mass or infiltration
* Concurrent local radiotherapy for potential or actual organ dysfunction by localized lymphoma mass or infiltration allowed

Surgery:

* Not specified

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2001-02

PRIMARY OUTCOMES:
Event-free survival

SECONDARY OUTCOMES:
Complete response
Overall survival
Disease-free interval
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Sonneveld, MD, PhD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (13):
- Netherlands (13):
  - Meander Medisch Centrum, Amersfoort
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Sint Antonius Ziekenhuis, Nieuwegein
  - Daniel Den Hoed Cancer Center at Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis - Locatie Leyenburg, The Hague
  - University Medical Center Utrecht, Utrecht
  - Isala Klinieken - locatie Sophia, Zwolle